CLINICAL TRIAL: NCT02677519
Title: A 12-Month Open Label Safety Study of Methylphenidate Hydrochloride Extended-Release Capsules (Aptensio XR®) in Children Ages 4-5 Years Diagnosed With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A 12-Month Open Label Safety Study of Aptensio XR® in Children Ages 4-5 Years Diagnosed With ADHD
Acronym: EF004
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-BP-EF004
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; children; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 10 mg Aptensio XR (Experimental): 10 mg methylphenidate, extended release
  Interventions: Drug: Aptensio XR
- 15 mg Aptensio XR (Experimental): 15 mg methylphenidate, extended release
  Interventions: Drug: Aptensio XR
- 20 mg Aptensio XR (Experimental): 20 mg methylphenidate, extended release once daily
  Interventions: Drug: Aptensio XR
- 30 mg Aptensio XR (Experimental): 30 mg methylphenidate, extended release
  Interventions: Drug: Aptensio XR
- 40 mg Aptensio XR (Experimental): 40 mg methylphenidate, extended release
  Interventions: Drug: Aptensio XR
- 50 mg Aptensio XR (Experimental): 50 mg methylphenidate, extended release
  Interventions: Drug: Aptensio XR
- 60 mg Aptensio XR (Experimental): 60 mg methylphenidate, extended release
  Interventions: Drug: Aptensio XR

INTERVENTIONS:
Drug: Aptensio XR — Orally-administered extended release formulation of methylphenidate; once daily dosing
  Other Names: Methylphenidate Extended Release

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of methylphenidate hydrochloride extended-release capsules (Aptensio XR®) in children aged 4-5 years who have been diagnosed with attention-deficit/hyperactivity disorder (ADHD).

Safety and tolerability will be evaluated by assessing treatment-emergent adverse events (TEAEs) blood pressure, pulse, height, weight, electrocardiograms (ECGs), laboratory The primary objective of this study is to evaluate the long-term (12-month) safety and tolerability of Aptensio XR® in children aged 4 to less than 6 years who have been diagnosed with ADHD.

Safety and tolerability will be evaluated by assessing treatment-emergent adverse events (TEAEs) blood pressure, pulse, height, weight, electrocardiograms (ECGs), laboratory values and Columbia Suicide Severity Rating Scale (C-SSRS). Disturbances in sleep (quantity and quality) patterns will also be assessed using the Child Sleep Habits Questionnaire (CSHQ).

Secondary objectives include assessment of long-term efficacy of Aptensio XR®.

Secondary measures include:

* Investigator administered Attention-Deficit/Hyperactivity Disorder Rating Scale Preschool Version (ADHD-RS-IV Preschool Version)
* Clinical Global Impressions-Severity Scale (CGI-S )
* Connors Early Childhood Behavior-Parent Short form [Conners EC BEH-P(S)]

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 4 to less than 6 years inclusive at the time consent was given to participate in Prior Studies. New Subjects must be at least 4 years but less than 6 years of age when written consent is given to participate in this trial.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | 12 month maintenance phase
  Incidence of TEAEs during maintenance phase
Columbia Suicide Severity Rating Scale (C-SSRS) | 12 month maintenance phase
  Standardized assessment of suicide risk
Vital signs | 12 month maintenance phase
  blood pressure, pulse, height, weight
12-lead electrocardiogram | 12 month maintenance phase

SECONDARY OUTCOMES:
ADHD-RS-IV Preschool Version | 12 month maintenance phase
  Investigator administered Attention-Deficit/Hyperactivity Disorder Rating Scale Preschool Version (ADHD-RS-IV Preschool Version) to assess ADHD severity and functioning
Clinical Global Impressions-Severity Scale (CGI-S) | 12 month maintenance phase
  This scale provides a global rating of illness severity and improvement during the study. The subject is rated relative to the clinician's past experience with other patients who have the same diagnosis. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (among the most severely ill patients).
Connors Early Childhood Behavior-Parent Short [ConnorsEC BEH-P(S)] | 12 month maintenance phase
  Assesses behavior of preschool-aged children 2 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Center for Psychiatry And Behavioral Medicine Inc.; Scott Kollins, MD, Principal Investigator — Department of Psychiatry & Behavioral Sciences, Duke University, Durham, NC
Locations (2):
- United States (2):
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Childress AC, Foehl HC, Newcorn JH, Faraone SV, Levinson B, Adjei AL. Long-Term Treatment With Extended-Release Methylphenidate Treatment in Children Aged 4 to <6 Years. J Am Acad Child Adolesc Psychiatry. 2022 Jan;61(1):80-92. doi: 10.1016/j.jaac.2021.03.019. Epub 2021 Apr 20. PMID 33892111